CLINICAL TRIAL: NCT07359508
Title: Effect of Desflurane v/s Propofol on the Optic Nerve Sheath Diameter in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Desflurane v/s Propofol on the Optic Nerve Sheath Diameter
Acronym: ONSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: All India Institute of Medical Sciences, Raebareli, UP (Unknown)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, Vijay, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2; AllMS (Other: AIIMS Raebareli)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Propofol Target-controlled Infusion; Desflurane; Optic Nerve Sheath Diameter
Keywords: propofol; ONSD
MeSH Terms: interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Experimental): propofol infusion will be given in this group after induction of the patient
  Interventions: Drug: Propofol (Group P)
- Desflurane (Experimental): desflurane inhalation will be given in this group, after induction
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — In the D group, anesthesia was maintained with oxygen/air (40:60), desflurane, fentanyl and vecuronium
  Arms: Desflurane
Drug: Propofol (Group P) — In the P group, anesthesia was maintained with oxygen/air (40:60), propofol infusion @50 to 100mcg/kg/min, fentanyl and Vecuronium
  Arms: Propofol group

SUMMARY:
effect of propofol vs desflurane on ONSD

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-60 years ASA grade I or II scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* patients with ophthalmological and cerebrovascular diseases, systemic infections, psychiatric disorders, pregnancy, Intracranial space occupying lesion, abnormal liver/kidney functions prior myocardial infarction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter(ONSD) | before induction, introperative period for every 10 minutes
  ONSD will be measured in the operation thetaer

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS, Raebareli, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol